CLINICAL TRIAL: NCT06012331
Title: Clinical and Radiographic Evaluation of Revascularization of Immature Anterior Permanent Teeth Using (CGF) Versus (BC)
Brief Title: Clinical and Radiographic Evaluation of Revascularization of Immature Anterior Permanent Teeth Using Concentrated Growth Factor (CGF) Versus Blood Clot (BC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hana Ahmed Omer, PhD researcher in pediatric dentistry and public health department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: dental pulp revascularization
Record Dates: First submitted 2023-08-07; First posted 2023-08-25 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-09

CONDITIONS: Revascularization
MeSH Terms: interventions — Blood Coagulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentrated Growth Factor (CGF) (Experimental): Concentrated growth factor (CGF) is relatively a new generation of platelet concentrate product, it contains more cytokines and growth factors compared with PRP and PRF also promotes the proliferation, migration, and differentiation of stem cells
  Interventions: Procedure: concentrated growth factors in open apex; Procedure: Blood Clot (BC)
- Blood Clot (BC) (Active Comparator): Inducing bleeding to facilitate healing is a common surgical procedure. The blood clot formed after hemorrhage, acts as a scaffold and rich source of growth factors, and could play an important role in tissue repair in the canal. The growth factors could stimulate differentiation, growth, and maturation of fibroblasts, odontoblasts and cementoblasts, from the immature undifferentiated mesenchymal cells in the newly formed tissue matrix
  Interventions: Procedure: concentrated growth factors in open apex; Procedure: Blood Clot (BC)

INTERVENTIONS:
Procedure: concentrated growth factors in open apex — Dry canals with paper points. A 10 ml of venous blood will be collected and transferred to sterile tubes without anticoagulant solutions by a trained nurse. The tubes will be centrifuged machine using a one-step centrifugation protocol at variable rpm, after centrifugation, four layers will be obtained: the first layer at the top is serum, second layer is the fibrin buffy coat, the third layer is the liquid phase containing growth factors, The concentrated growth factor was separated from the red blood cells and serum using sterile scissors.
  CGF will be packed into canal to the full working length using sterile pluggers.
  The coronal level of the CGF gel is near the cervical area above cementoenamel junction and white MTA placed as capping material after CGF, then GIC and composite restoration
Procedure: Blood Clot (BC) — 1. Create bleeding into the canal by over-instrumenting (induce by rotating a pre-curved K-file at 2 mm past the apical foramen with the goal of having the entire canal filled with blood to CEJ level)
  2. Stop bleeding at a level that allows for 3-4 mm of restorative material.
  3. Then white MTA as a coronal plug material be followed by GIC, then composite restoration.

SUMMARY:
The aim of this study is to compare clinical and radiographic evaluation treatment of necrotic immature permanent teeth using:

1. Concentrated Growth Factor
2. Blood Clot

DETAILED DESCRIPTION:
Rationale for conducting the research:

Concentrated growth factor (CGF) is relatively a new generation of platelet concentrate product, it contains more cytokines and growth factors compared with PRP and PRF also promotes the proliferation, migration, and differentiation of stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 8_14 years.
2. Anterior tooth diagnosed with necrotic pulp (due to trauma, caries, or anomaly) responded negatively to sensibility tests.
3. Teeth not indicated for post and core.
4. A cooperative and compliant patient/parent.
5. Patients not allergic to medicaments necessary to complete the procedure.
6. Patients with no history of chronic systemic diseases.

Exclusion Criteria:

1. Medically compromised patient.
2. Teeth with vertical fractures.
3. Non-restorable teeth.
4. Teeth when bleeding could not be induced.
5. Unable to attend follow-up visits.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
clinically successful treatment | 3,6,9,12 months
  The treatment will be considered to be clinically successful when. Absence of pain will record it by verbal question to patient/ parent. Absence of tenderness to percussion) will record it by percussion test (by the back of the dental mirror) Absence of swelling and fistula or sinus tract -- will record it by visual clinical examination

SECONDARY OUTCOMES:
Radiographic Success treatment | 6, 12 months
  The treatment will be considered to be Radiographic Success when.
  * Root elongation (increased root length): will be assessed in mm through a radiographic x-ray system measure from cementoenamel junction to the apex.
  * Root maturation: increased root dentin thickness will be assessed in mm through a radiographic x-ray system for each case and will be calculated as the difference between the outer root area and the pulp space area.
  * Absence or reduce in the size of periapical radiolucency: will be assessed in mm through a radiographic x-ray system.

REFERENCES:
- [Background] Kasprisin DO, Heiss R, Rausen AR. Cholelithiasis during remission of acute lymphocytic leukemia in a child. Clin Pediatr (Phila). 1981 Oct;20(10):678. No abstract available. PMID 6944166
- [Background] Ruskin KJ, Tissot M. A new method of communication between anesthesiologists. Anesthesiology. 1993 Oct;79(4):867. doi: 10.1097/00000542-199310000-00037. No abstract available. PMID 8214771